CLINICAL TRIAL: NCT04923178
Title: A Multi-Center Natural History of Urothelial Cancer and Rare Genitourinary Tract Malignancies
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000302; 000302-C
Record Dates: First submitted 2021-06-10; First posted 2021-06-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-21

CONDITIONS: Urothelial Cancer; Bladder Cancer; Genitourinary Cancer; Urogenital Neoplasms; Urogenital Cancer
Keywords: bladder/urachal adenocarcinoma; renal tumors; penile cancers; small cell neuroendocrine carcinoma of the prostate; Renal Cell Carcinoma; Natural History
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urogenital Neoplasms; Urachal adenocarcinoma; Carcinoma, Renal Cell; Penile Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1 / Urothelial cancer: Participants with urothelial cancer.
- 2 / Rare Bladder or Urinary Tract Histology: Participants with small cell carcinoma, adenocarcinoma, urachal squamous cell carcinoma, or pure sarcomatoid carcinoma. These pure histologies can occur in the bladder and/or urinary tract.
- 3 / Urothelial Carcinoma Variants: Participants diagnosed with a urothelial variant histologies at any stage.
- 4 / Rare GU Tumors: Participants with renal medullary carcinoma, testicular Sertoli or Leydig cell tumors, penile cancer, refractory germ cell tumors.

SUMMARY:
Background:

Tumors in the genitourinary tracts can occur in the kidney, bladder, prostate, and testicles and can have common and rare histologies. Some cancers that occur along the genitourinary (GU) tract are rare. Some GU tumors are so rare that they are not included in treatment studies or tissue banks. This makes it hard for researchers to determine standards of care. Researchers want to learn more about common and rare GU tumors.

Objective:

To learn more about urinary tract cancers.

Eligibility:

People ages 18 and older with urinary tract or GU cancer such as bladder, kidney, testicular, prostate, penis, or neuroendocrine cancer.

Design:

Participants will be screened with questions about their medical history. Their medical records will be reviewed.

Participants will have a physical exam. They will give blood and urine samples. They will complete a survey about their family cancer history. Clinical photographs will be taken to document skin lesions.

Participants may have imaging scans of their chest, abdomen, and pelvis. They may have a contrast agent injected into their arm.

Participants will get recommendations about how to best manage and treat their cancer. They can ask as many questions as they would like.

Participants will provide existing tumor samples if available. They may have optional tumor biopsies up to twice a year. For needle biopsies, the biopsy area will be numbed and they will get a sedative. A needle will be inserted through their skin to collect a tumor sample. For skin biopsies, their skin will be numbed. A small circle of skin will be removed.

Some blood and tumor samples may be used for genetic tests.

Participants will have frequent follow-up visits. If they cannot visit NIH, their home doctor will be contacted. They will be followed on this study for life....

DETAILED DESCRIPTION:
Background:

* Histological variants of the genitourinary (GU) tract include bladder/urachal adenocarcinoma, squamous cell carcinoma, and small cell carcinoma; variants of urothelial carcinoma including plasmacytoid, sarcomatoid; renal tumors including sarcomatoid renal cell carcinoma and renal medullary carcinoma; penile cancers; micropapillary, giant cell, lipid rich, clear cell and nested variants, large cell neuroendocrine carcinoma, lymphoepithelioma-like carcinoma and mixed patterns; small cell neuroendocrine carcinoma of the prostate, testicular Sertoli or Leydig cell tumors, and papillary and chromophobe renal cell carcinoma (RCC).
* Some GU tumors occur so infrequently that they are not systematically captured by currently available registries, treatment protocols, or tissue banks. The rarity of these tumors limits the sufficient numbers of patients needed in larger randomized clinical studies to characterize standard treatments or disease course.
* Systematic and longitudinal collection and annotation of clinical history, tissue samples, imaging studies, and other pertinent information in participants with these rare tumors will yield future knowledge and help with the development of subsequent prospective studies to optimize diagnosis and treatment paradigms for less common GU tumors.

Objective:

-Characterization of the natural history of urothelial and GU tract malignancies.

Eligibility:

-Participants >= 18 years of age diagnosed with urothelial or GU tract malignancies.

Design:

* This will be a long-term multi-center study to comprehensively study participants with GU tumors.
* Medical history will be collected, and participants followed throughout the course of their illnesses, with particular attention to patterns of disease presentation, recurrence and progression, response to therapies, and duration of responses.
* Tissue samples and blood will be obtained from participants during this study.
* A broad spectrum of scientific experiments, including genomics and immune monitoring will be performed.
* We anticipate accruing 1000 participants on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed urothelial or rare genitourinary cancer including but not limited to the following: small cell carcinoma of the bladder; adenocarcinoma of the bladder; squamous cell carcinoma of the bladder; plasmacytoid urothelial carcinoma; any penile cancer; any testicular cancer, sarcomatoid renal cell carcinoma; sarcomatoid urothelial carcinoma; renal medullary carcinoma or other miscellaneous histologic variants of the urothelial carcinoma, such as, but not limited to micropapillary, giant cell, lipid-rich, clear cell and nested variants, large cell neuroendocrine carcinoma, lymphoepithelioma-like carcinoma and mixed patterns will be considered, as well as small cell neuroendocrine prostate cancer, testicular Sertoli or Leydig cell tumors. Any genitourinary cancer can be included at the principal investigator's discretion.
* Age >=18 years.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2041-12-01 (Estimated); Study Completion 2042-12-01 (Estimated)

PRIMARY OUTCOMES:
natural history of urothelial and rare genitourinary cancer | ongoing
  clinical presentation, patterns of disease progression, therapeutic response, disease recurrence and participant overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000302-C.html